CLINICAL TRIAL: NCT01677819
Title: Inhibition Control of Children and Adolescents With Attention-Deficit/Hyperactivity Disorder
Brief Title: Inhibition Control of Children and Adolescents With ADHD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Susan Shur-Fen Gau, National Taiwan University Hospital
Other Study IDs: 201109027RD
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objectives of this study are to investigate:

1. the effect of methylphenidate on attention;
2. the relations between methylphenidate and inhibition control and working memory;
3. the relations between inhibition control and verbal attention and working memory;
4. the effect of methylphenidate on the changes of neuropsychological functioning and blood pressure.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD), characterized by inattention, hyperactivity and impulsivity, is an early onset, highly heritable, clinically heterogeneous, long-term impairing disorder with tremendous impact on individuals, families, and societies. It affects 5-10% of school-aged children worldwide (7.5% in Taiwan). Methylphenidate, a stimulant, is effective in treating these patients. Studies in Taiwan show no effect of methylphenidate on blood pressure. There are evidences show that the change of blood pressure was associated with inhibition of impulsive behaviors. Stop Signal Task(SST) is used to assess the improve of inhibition control after methylphenidate response. By using repeated outcome measurements, we anticipate that this study will evaluate the improvement of neuropsychological performances after medication and determinie the association between medication response and neuropsychological functions and vital signs in a Taiwanese sample.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the subjects are (1)that subjects have a clinical diagnosis of ADHD defined by the DSM-IV which was made by a full-time board-certificated child psychiatrist; (2)their ages range from 10 to 18 when we conduct the study; (3)their IQ greater than 80; and (4)they are under treatment of methylphenidate.

Exclusion Criteria:

The subjects will be excluded from the study if they currently meet criteria or have a history of the following condition as defined by DSM-IV: Schizophrenia, Schizoaffective Disorder, Organic Psychosis, or Pervasive Developmental Disorder.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We will recruit 60 children and adolescents, aged 10 to 18, who are diagnosed with ADHD at the Department of Psychiatry, National Taiwan University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-11; Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan